CLINICAL TRIAL: NCT06745349
Title: The Sleep Course: Examining the Feasibility, Acceptability, and Effectiveness of an Online Sleep Intervention for Adults With Self-reported Sleep Difficulties
Brief Title: The Sleep Course: An Online Sleep Intervention for Adults With Self-reported Sleep Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 873
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Insomnia; Depression; Anxiety
Keywords: Internet; Internet-Delivered CBT; Digital Mental Health Interventions; Insomnia; Sleep Difficulties; Depression; Anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICBT for insomnia (Experimental): Therapist-guided, Internet-delivered cognitive behavioral therapy for insomnia (ICBTi)
  Interventions: Behavioral: Sleep Course

INTERVENTIONS:
Behavioral: Sleep Course — The Sleep Course previously developed and evaluated in Australia will be delivered to clients meeting participation criteria. The Sleep Course is four lessons long and is offered with once weekly therapist support for 8 weeks where clients are encouraged to email the assigned therapist for support each week. The therapist reviews client progress in the Course and emails clients once per week on a designated check in date. Sometimes the therapist will call the client. Phone calls are typically made if a client is not logging in or if the therapist feels that a phone call would be a helpful way to provide support.

SUMMARY:
This study evaluates an internet-delivered cognitive behavioural therapy for insomnia (ICBTi) intervention, known as the Sleep Course, within a routine online therapy clinic (the Online Therapy Unit). The Sleep Course will specifically be offered to clients with self-reported sleep difficulties (i.e., falling or staying asleep or waking early) and daytime distress and or impairment. This study aims to replicate the effectiveness and acceptability of the previously evaluated Sleep Course when delivered in Australia. The investigators will also assess uptake and completion rates within the clinic as well as demographic and clinical characteristics of individuals enrolled in the Sleep Course.

DETAILED DESCRIPTION:
To improve access to effective psychological treatment, Internet-delivered Cognitive Behaviour Therapy (ICBT) has been developed. ICBT delivers therapeutic content via structured online lessons usually over several months, teaching the same skills that are taught in face-to-face cognitive behaviour therapy. In routine practice, ICBT is often accompanied by brief therapist support offered via secure messaging and/or phone calls. A growing body of research supports the effectiveness of ICBT for a variety of conditions, including depression, anxiety, alcohol misuse, and insomnia. For insomnia, ICBTi has been shown to result in improvements on various sleep measures, comorbid anxiety and depression, and quality of life, with outcomes comparable to face-to-face treatment.

Importantly, there are a growing number of studies showing the effectiveness of ICBT for depression and anxiety extends to routine care. However, there are fewer studies exploring ICBTi in routine care, particularly when minimal exclusion criteria are imposed. This research is important because sleep difficulties and insomnia are common, distressing and often disabling and frequently comorbid with mood or anxiety disorders as well as various physical conditions. Moreover, access to specialized psychological services, such as CBTi, is often limited, despite CBTi being a well-established first-line treatment, which many clients find more acceptable than medication. Two key aspects of CBTi are stimulus control and sleep restriction though other strategies such as cognitive restructuring and relaxation are also commonly included. ICBTi offers a promising approach for expanding access to evidence-based treatment for insomnia. This is especially critical given the high personal and societal costs of leaving insomnia untreated.

From past research, the investigators have found that approximately 73% of clients enrolled in the routine clinic that offers ICBT for anxiety and depression also reported significant sleep problems. Of these, only 30% accessed an additional sleep resource to address their sleep concerns. While improvements in sleep were observed among all clients enrolled in ICBT, average post-test treatment scores indicated many clients still had significant difficulties with insomnia. In another study conducted within the investigators' Unit, the investigators explored whether offering an insomnia-focussed lesson at the beginning of ICBT would improve insomnia symptoms. In this study, the investigators found that clients experienced large reductions in insomnia symptoms at a faster rate than when clients did not receive the insomnia lesson at the beginning of ICBT. However, even with these improvements, many clients continued to report clinically significant levels of insomnia post-treatment, indicating that further support for insomnia symptoms may be beneficial.

Overall, given that the investigators ICBT program does not appear to be fully meeting the sleep needs of clients who have depression and anxiety, as well as the needs of clients who have sleep problems or insomnia and do not want ICBT for depression and anxiety, the investigators believe it would be valuable to explore the benefits of offering ICBTi in the routine care clinic. This is especially important for routine care settings where inclusivity is key and services should be broadly accessible.

One such program that shows promise among clients with diverse sleep difficulties is the Sleep Course. The current study therefore aims to explore the extent to which this ICBTi program will be used by clients seeking services within the routine online clinic. Additionally, the study will explore the demographic and clinical characteristics of clients who seek ICBTi, as well as the acceptability and effectiveness of the ICBTi program. The data collected will shape long-term practices within the Online Therapy Unit and has potential to significantly enhance service delivery. The research will also provide valuable insights for other online clinics regarding the potential of offering ICBTi in routine online care. By exploring the program's use, client characteristics, acceptability, and effectiveness, this study will contribute to a broader understanding of how ICBTi can be successfully integrated into routine online services, ultimately improving access to evidence-based treatment for insomnia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Living in Saskatchewan for the treatment period;
* Self-reported difficulty with sleep (i.e., difficulty falling, staying asleep or waking up early) causing daytime distress and or impairment;
* Has comfort using and access to a device or computer with Internet in a private location;
* Read and understand English;
* Consent to Sleep Course, online therapy as provided by Unit, and associated research.

Exclusion Criteria:

* Current severe medical or psychiatric disorder that requires immediate or alternate treatment (e.g. current and recent mania or psychosis requiring hospitalization, actively suicidal and unable to keep themselves safe, medical condition requiring immediate surgery or other invasive treatment, severe substance use);
* Taking part in another treatment at our clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia symptoms | Screening, weeks 1, 2, 3, 4, 5, 6, 7 (post-treatment), and 3-month follow-up
  Insomnia Severity Index (ISI). Includes 7 items rated on a 0 to 4 scale. Higher total scores indicate greater severity of insomnia symptoms over the past two weeks. Scores range from 0 to 28.

SECONDARY OUTCOMES:
Change in sleep diary scores | Baseline and week 7 (post treatment)
  The core Consensus Sleep Diary (CSD) consisting of 9 items, will be administered to clients each morning for 7 consecutive days, asking about their sleep the previous night. Participants will record the time they went to bed, time to initiate sleep, time they woke up in the morning, time of final awakening, and time they got out of bed in the morning (in clock). Participants will also record the number (in numbers) and duration of awakenings during the night (in minutes). Using a 6-point Likert scale ranging from 0 to 5, participants will indicate the quality of their sleep with higher scores indicating more restorative sleep quality. An additional open-ended item is added for comments. Two extra questions on napping-extracted from the Expanded Consensus Sleep Diary for Morning- will be included. Using this, participants will record if they napped the previous day (yes/no), and for how long (in minutes). There is no overall score for the scale, each parameter is analyzed separately.
Change in sleep quality | Screening, week 7 (post treatment) and 3-month follow-up
  Pittsburgh Sleep Quality Index (PSQI). A 19-item survey rated on a 0 to 3-point scale. This survey is used to assess sleep dysfunction over the past month and produces scores for subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, use of medication, daytime dysfunction, and higher scores indicate severe difficulties in each area. A sum of the scores from these factors produces a global score between 0-21, where higher global scores indicate more severe sleep disturbances.
Change in sleep quality | Weeks 1, 2, 3, 4, 5, and 6
  Pittsburgh Sleep Quality Index (PSQI- 4 Items). A 4-item survey that assesses quality of sleep. Items on this scale are measured on a 4-point Likert scale ranging from 0-3, and scores range from 0-12, with higher scores indicating worse sleep quality. This measure is used by clinicians to monitor client sleep.
Change in attitudes and beliefs about sleep | Screening, week 7 (post-treatment) and 3-month follow-up
  Dysfunctional Beliefs and Attitudes about Sleep- 16 item (DBAS-16) with items rated on a 0 to 10-point scale. Scores range from 0 to 160 with higher scores indicating greater dysfunctional beliefs about sleep.
Change in depression | Screening, week7 (post treatment) and 3-month follow-up
  Patient Health Questionnaire - 9 Item (PHQ-9). Includes 9 items rated 0 to 3. Higher total scores indicate greater severity of depression. Scores range from 0 to 27. Clinical cutoff of ≥10 indicate clinically significant depression.
Change in depression and anxiety | Weeks 1, 2, 3, 4, 5, and 6
  Patient Health Questionnaire - 4 Item (PHQ-4) involves rating 4 items on a scale from 0 to 3, with scores ranging from 0 to 12. Higher total scores indicate greater severity of depression and anxiety symptoms. Additionally, item #9 of the PHQ-9 is presented alongside the PHQ-4 to monitor client's wellbeing. This item is rated on a scale from 0 to 3, with higher scores indicating more severe self-harm or suicidal ideology. However, the score from this item is not included in the overall PHQ-4 score. This measure is used by clinicians to monitor client's mental health symptoms.
Change in anxiety | Screening, week 7 (post treatment) and 3-month follow-up
  Generalized Anxiety Disorder - 7 Item (GAD-7). Includes 7-items used to assess generalized anxiety disorder. Items are rated on a 0 to 3-point Likert scale. Total score range from 0 to 21, and higher total scores indicate greater severity of anxiety. Clinical cutoff of ≥10 indicates clinically significant anxiety.
Lesson reflection | Weeks 2, 3, 4, 5, 6, and 7 (post treatment)
  Lesson reflection questionnaire - A bespoke 6-item survey that inquires about which lesson and resources clients worked on, effort, understanding, helpfulness, and client successes and challenges over the previous week. This survey is used for clinicians to monitor treatment. No score is calculated or created.
Evaluation of treatment | Week 7 (post treatment)
  Treatment Satisfaction Survey. A bespoke questionnaire consisting of 15 items with varying response formats measuring treatment satisfaction. The questionnaire utilizes a combination of Likert-scale (5-point (0-4)and 6-point (0-5) ), open-ended, and dichotomous yes/no response options to gauge participants' perception of the course. No overall score is calculated or reported for this questionnaire.
Engagement | Collects engagement from time of consent to 3 month follow-up
  The system collects information on number of lessons completed, number of additional resources accessed, number of emails sent to and received from therapist. Participants' engagement is calculated by averaging the sum from all of the components listed above.
Background Information | Screening
  Background information including demographic questions will be collected at screening for descriptive purposes. No scores are calculated.
Sleep history & treatment history | Screening
  Sleep and treatment history questions will be administered at screening for descriptive purposes. No scores are calculated based on these questions.

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Helpful Links Provided by University of Regina — https://www.onlinetherapyuser.ca/